CLINICAL TRIAL: NCT06736249
Title: Attivazione Farmacologica Di HIF-1α Come Nuovo Approccio Terapeutico Per Contrastare La Perdita Di Fibre Glicolitiche in Pazienti Sarcopenici.
Brief Title: HIF-1α Stabilization As a Novel Therapeutical Approach for Sarcopenia.
Acronym: HIF2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HIF2
Record Dates: First submitted 2024-01-16; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sarcopenic group (Experimental): This group will undergo a DXA total body to confirm sarcopenia
  Interventions: Diagnostic Test: Sarcopenic group; Other: Muscle harvesting
- Control (Other): This group is a control group of young active patients to compare with the sarcopenic group
  Interventions: Other: Muscle harvesting

INTERVENTIONS:
Diagnostic Test: Sarcopenic group — The sarcopenic group will undergo a DXA total body to define the sarcopenic stage.
  Arms: Sarcopenic group
Other: Muscle harvesting — A piece of discarded muscle during surgery will be collected

SUMMARY:
Age-related sarcopenia is associated with reduced mobility, functional decline and disability, falls, and mortality in the elderly. Loss of skeletal muscle is the focus of the disease and is the result of progressive atrophy and loss of glycolytic-type muscle fibers. Muscle mass declines at a rate of 3-5% per decade after thirty years, and the decrease accelerates further after sixty years (Patel et al., 2013). As life expectancy increases worldwide, it is clear that sarcopenia is considered a major contributor to healthcare costs and that even a small reduction in the prevalence of sarcopenia could result in substantial savings in healthcare resources (Goates et al., 2019). In this context, the present proposal aims to develop a new therapeutic approach based on the activation of HIF-1alpha, which has been shown to promote skeletal muscle hypertrophy, to prevent and counteract sarcopenia, thereby reducing disability in the elderly and the impact on the national health care system.

DETAILED DESCRIPTION:
The crucial role played by hypoxia-inducible factor-1α (HIF-1α) during myogenesis has been demonstrated in two recent publications by the proponent group (Cirillo et al., 2017a;Cirillo et al., 2020). Specifically, it was shown that proliferating murine myoblasts treated for 24 hours under 1% O2 (hypoxia) conditions in growth medium and then stimulated to differentiate for 7 days under normoxic conditions (21% O2) showed the formation of hypertrophic myotubes with a 1.4-fold increase in differentiation index compared with normoxic controls. These results were confirmed by analysis of key differentiation markers. Specifically, hypoxic pretreated myoblasts showed a 3-, 2.4-, and 1.33-fold increase in MyoD nuclear localization, myogenin expression after 3 days of differentiation, and MHC expression at the end of the differentiation process compared with controls, respectively. Moreover, we confirmed these findings in skeletal muscle biopsies from elderly sarcopenic patients compared with those from young individuals. We found a decrease in the expression of HIF-1α and its target genes in sarcopenia, as well as of PAX7, the major stem cell marker of satellite cells, whereas the atrophy marker MURF1 was increased. We also isolated satellite cells from muscle biopsies and cultured them in vitro. We found that a pharmacological activation of HIF-1α and its target genes caused a reduction in skeletal muscle atrophy and activation of PAX7 gene expression. In conclusion, in this work we found that HIF-1α plays a role in sarcopenia and is involved in satellite cell homeostasis (Cirillo et al., 2022).

Considering our preliminary data, the first part of our project will focus on patient recruitment and clinical characterization. Specifically, analyzes will be performed on two separate groups: the sarcopenic group, consisting of 60 patients affected by sarcopenia according to the most recent guidelines (> 65 years), and the control group, consisting of 45 patients who are not sarcopenic (aged between 18 and 35 years). The study will be conducted according to the rules of the hospital ethics committee and patients will be required to sign an informed consent form to participate in the study. Patients will be recruited for 24 months, with 6 months available for data analysis. Recruitment will take place during routine orthopedic examinations at the IRCCS Istituto Ortopedico Galeazzi in patients scheduled for orthopedic surgery (hip replacement due to osteoarthritis, proximal femur fractures, and ALC reconstructive surgery). Patients with comorbidities, including obesity-related sarcopenia and diabetes, will be excluded from the study. All patients will undergo to (a) DXA total body, which allows quantification of the three body components bone mineral, fat, and bone mineral-free mass, (b) hand-held dynamometry to assess grip strength, and (c) anthropometric analysis (BMI) to estimate body fat. A blood sample will be collected to determine the extent of sarcopenia by serological analysis. This involves measuring amino-terminal pro-peptide of procollagen type III (P3NP), c-terminal agrin fragment 22 (CAF22), osteonectin, irisin, fatty acid binding protein 3 (FABP3), and macrophage migration inhibitory factor (MIF), which are considered the main candidate biomarkers of sarcopenia (Nogueira et al., 2019;Qaisar et al., 2020). Following patient recruitment, the study will aim to identify changes in HIF-1alpha signaling during sarcopenia. Specifically, multiple skeletal muscle biopsies, normally discarded during surgery, will be collected from sarcopenic and control groups to set up multi-omics approaches and histological assays. In particular, total proteins will be extracted by skeletal muscle sample to perform proteome analyzes based on mass spectrometry and cellular bioenergetic metabolism assay using Seahorse Real-Time Cell Metabolic Analysis in our laboratory. Statistical analysis of the proteome and metabolome data will focus on changes in cross-talk between HIF signaling and mitochondrial activity. The proteome results will be technically validated by a Western blot approach using specific antibodies. Only the proteins showing a true difference in expression of at least 0.6 will be considered. On the other hand, skeletal muscle biopsies will also be used for histological examination. The main focus will be on 1) activation of satellite cells by the specific antibody PAX7, 2) quantification of skeletal muscle atrophy by the specific antibody MuRF1, 2) and changes in muscle fiber composition using specific antibodies directed against myosin heavy chain type I, IIA, and IIB.

ELIGIBILITY:
Inclusion Criteria:

* For non-sarcopenic patients aged 18 to 35 years, for sarcopenic patients aged > 65 years.
* 18 ≤ body mass index (BMI) ≤ 30 kg/m2.
* For the sarcopenic group:

  1. non-inflammatory degenerative joint disease, including osteoarthritis and outcomes of congenital hip dysplasia.
  2. surgeries to correct hip joint deformities
  3. fractures of the proximal femur involving the head that cannot be treated with reduction and fixation techniques
  4. hip revision surgery.
* For the non-sarcopenic group:

  5. traumatic injury to the anterior cruciate ligament.

Exclusion Criteria:

* Use of medications that may affect metabolism or bone,
* Signs of diseases known to affect muscle-bone metabolism.
* Bone metastases or disease at the surgical site.
* Positive for HCV, HIV, HBV, or TPHA.
* Presence of infection or suspected hip infection.
* Inability to provide informed consent.
* Obesity (BMI ≥30kg/m2).
* Inability to undergo DXA total body in sarcopenic patients due to medical contraindications or claustrophobia.

For sarcopenic group: ASMI >7.0 kg/m2 form men and >5.5 kg/m2 for women; FMI <6 for men and <9 for women For control group: pregnancy or breastfeeding

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2023-05-25 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate that the pharmacological activation of HIF-1alpha is an effective approach to counteract sarcopenia. | 18 months
  Satellite cells harvested from sarcopenic patients will be treated with FG-4592, a PHD inhibitor.At the end of the treatment, metabolic changes will be analyzed using Seahorse Real-Time Cell Metabolic Analysis.

SECONDARY OUTCOMES:
To perform a proteome analysis on the samples | 12 months
  Mass spectrometry and Western blot analysis
To evaluate metabolic differences between sarcopenic and control goups | 12 months
  Samples will be analyzed with Seahorse Real-Time Cell Metabolic Analysis

CONTACTS AND LOCATIONS:
Overall Officials: Laura Mangiavini, Principal Investigator — University of Milan, IRCCS Ospedale Galeazzi-Sant'Ambrogio
Locations (1):
- IRCCS Ospedale Galeazzi-Sant'Ambrogio, Milan, Europe, Italy

IPD SHARING:
Plan to Share IPD: No